CLINICAL TRIAL: NCT04347135
Title: Pilot Study Evaluating Endometriosis With 16α-(18)F-fluoro-17β-estradiol ([F-18] FES) PET/MRI
Brief Title: Evaluating Endometriosis With 16α-(18)F-fluoro-17β-estradiol ([F-18] FES) PET/MRI
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No Enrollment
Sponsor: Annie (Annie) T. Packard (Other)
Responsible Party: Sponsor-Investigator, Annie (Annie) T. Packard, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-004345
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- F-18 FES PET/MRI (Experimental): 16α-(18)F-fluoro-17β-estradiol ([F-18] FES)
  Interventions: Drug: F-18 FES

INTERVENTIONS:
Drug: F-18 FES — F-18 FES PET/MRI for detection of endometriosis.

SUMMARY:
Researchers are trying to improve the detection of endometriosis using F-18 FES PET/MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

- Premenopausal women (18-50) with endometriosis

Exclusion Criteria:

* Postmenopausal women
* AP diameter when lying supine greater than 32 cm (too large for PET/MRI)
* Unable to undergo PET/MRI for any reason (metal implants, severe claustrophobia)
* Unable to receive IV Gadolinium contrast for any reason (renal failure eGFR < 60, contrast allergy)
* Pregnant (Urine test will be provided for all patients)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Detection of Endometriosis | 24 months
  Comparisons will be made descriptively between conventional MRI imaging, FES PET/MRI imaging and surgical/pathologic findings. Outcome data include number of detected lesions, differences in the accuracy for detection of active disease versus inactive fibrosis, and confidence score.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Packard, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials